CLINICAL TRIAL: NCT06756074
Title: Impact of Reinforced Pancreaticojejunostomy With or Without Tissue Adhesive Glue Modified Cyanoacrylate (Glubran 2) Following Pancreaticoduodenectomy, Randomized Controlled Clinical Trial.
Brief Title: Reinforced Pancreaticojejunostomy With or Without glubran2
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Saleh Khairy Saleh MD, Lecturer, Minia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1350/11/2024
Record Dates: First submitted 2024-12-24; First posted 2025-01-01 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Pancreatic Fistula; Pancreas Cancer; Periampullary Carcinoma; Pancreatic Ductal Adenocarcinoma
MeSH Terms: conditions — Pancreatic Fistula; Pancreatic Neoplasms | interventions — glubran 2; Pancreaticojejunostomy

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Masking Description: Surgeons are not blinded due to the intervention's nature; care provider , assessors, and analysts are blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Reinforced pancreaticojejunostomy with tissue adhesive glue modified cyanoacrylate (glubran 2) (Experimental): Reinforced pancreaticojejunostomy with tissue adhesive glue modified cyanoacrylate (glubran 2)
  Interventions: Drug: Reinforced pancreaticojejunostomy with tissue adhesive glue modified cyanoacrylate (glubran 2)
- Pancreaticojejunostomy without tissue adhesive glue modified cyanoacrylate (glubran 2) (Active Comparator): Pancreaticojejunostomy without tissue adhesive glue modified cyanoacrylate (glubran 2)
  Interventions: Procedure: Pancreaticojejunostomy without tissue adhesive glue modified cyanoacrylate (glubran 2)

INTERVENTIONS:
Drug: Reinforced pancreaticojejunostomy with tissue adhesive glue modified cyanoacrylate (glubran 2) — pancreaticojejunostomy was done with application of glubran 2: The blister pack was opened, and the sterile single-dose vial was released directly onto the operating table in a sterile environment, Draw the Glubran 2 out of the single-dose vial using a sterile syringe then put the syringe into applicator Glubran 2 was applied into anastomosis by applicator in spraying manner . Whenever possible, the area to be treated should be cleaned before application. When applied in such a minimal amount, once it had polymerized, Glubran 2 formed a thin adhesive layer. It was therefore essential not to apply more than one drop in the same point. A second layer of Glubran 2 may not be applied until the first had polymerized. Any excess product was removed using a dry swab within 5-6 seconds after application. Glubran 2 was not touched after application until the polymerization reaction is complete, as it may detach or not produce the desired effect.
  Arms: Reinforced pancreaticojejunostomy with tissue adhesive glue modified cyanoacrylate (glubran 2)
Procedure: Pancreaticojejunostomy without tissue adhesive glue modified cyanoacrylate (glubran 2) — Pancreaticojejunostomy without tissue adhesive glue modified cyanoacrylate (glubran 2)
  Arms: Pancreaticojejunostomy without tissue adhesive glue modified cyanoacrylate (glubran 2)

SUMMARY:
Pancreatic fistula is one of the most serious complication after pancreatoduodenectomy. To reduce pancreatic fistula, many authors recommend different techniques in pancreatojejunostomy. The purpose of this study is to determine which is the best method in preventing pancreatic fistula by enforce pancreaticojejunostomy with tissue glue and to investigate its long term clinical outcomes.

DETAILED DESCRIPTION:
Tissue adhesives have gained popularity in various fields of surgical practice. There are various types of tissue adhesives, each with their own adhesive mechanisms and uses. Basically, a tissue adhesive forms bonds with its substrate, ensuring sufficient adhesion. These bonds can either be chemical, of which covalent bonds are the strongest, or physical, including hydrogen bonds or van der Waals forces. Furthermore, the total strength of the glue bond depends on the balance between interaction within the tissue adhesive (cohesion) and between the tissue adhesive-substrate interface (adhesion). Tissue adhesives can either be glues, intended to independently connect various structures (i.e., wound edges), or sealants, used to cover and protect an anastomosis .

Except for external use, tissue adhesives can also be used intracorporeally. Various tissue adhesives are being used in cardiovascular surgery, plastic surgery, and, increasingly, surgery of the GI tract .

Tissue adhesives are promising tools for wound closure. They distribute forces throughout the wound more evenly and noninvasively than sutures and staples, are strong and flexible, and do not interfere with the wound-healing process. Also, the technique of tissue adhesive application to the wound is easy and standardizable, resulting in less variation in technique between surgeons .

By using tissue adhesives as sealants of GI anastomosis, enhancing standard anastomotic techniques. Numerous research projects have been undertaken to assess the applicability of available tissue adhesives in GI surgery; however, no recent literature provides the surgical community with an up-to-date overview of the progress in this field .

In addition to reducing the incidence of post operative pancreatic fistula, external pancreatic duct drainage may have other potential benefits, such as decreasing the length of hospital stay, reducing the need for additional interventions, and improving overall patient quality of life. However, these potential benefits must be weighed against the risks and drawbacks of external pancreatic duct drainage, including the potential for stent-related complications and the need for an additional procedure to remove the stent.

•After being informed about the study and potential risks, all patients giving written consent. Patients who meet the eligibility requirements will be randomized in a 1:1 ratio to external pancreatic drainage group and no external pancreatic drainage group.

ELIGIBILITY:
Inclusion Criteria:

* All the patients undergoing pancreaticoduodenectomy for cancer
* Patients able to give their informed consent

Exclusion Criteria:

* Unfit patients for surgery due to severe medical illness.
* Inoperable patients by imaging studies, irresectable tumors after laparotomy or diagnostic laparoscopy.
* Presence of distant metastasis .
* Patients refused to participate in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-01-15 (Actual); Primary Completion 2026-04-15 (Estimated); Study Completion 2026-05-15 (Estimated)

PRIMARY OUTCOMES:
the rate of Postoperative pancreatic fistula within 2 weeks after operation | within 2 weeks after operation
  Postoperative pancreatic fistula (POPF) is defined as a drain output of any measurable volume of fluid on or after postoperative day 3 with an amylase content greater than 3 times the serum amylase activity.

SECONDARY OUTCOMES:
Post-Pancreatectomy Hemorrhage | 90 days
  As defined by the International Study Group for Pancreatic Surgery (ISGPS), grade A, B and C rates
Delayed Gastric Emptying | 90 days
  As defined by ISGPS, grade A, B and C rates
Biliary fistula | 90 days
  Output of bile from drains on or by post operative day 3, pancreaticojejunostomy leak should be ruled out
Abdominal abscess | 90 days
  Collection >5cm in size, containing gas bubbles, determining systemic signs of infection
Acute pancreatitis | 1 day post index surgery
  Altered serum amylase count on post operative day 0 or 1
Wound infection | 90 days
  Superficial and Deep Surgical Site Incisional Infection as defined by the Center for Disease Control and Prevention
Blood transfusions | 90 days
  Need and number of packed red blood cells transfused
Reoperation | 90 days
  Need for new surgery due to severe morbidity
Readmission | 30 days after hospital discharge
  New admission within 30-days of discharge from hospital
Length of Hospital Stay | 1 year
  calculated from the day of surgery to the day of discharge, adding up the days after a possible re-admission
Mortality | 90 days
  Death related to surgical morbidity
Removal time of drain | From date of surgery until the date of the last drainage removal, whichever came first, assessed up to study completion, an average of 1 year
  The timing of removal of the drain tube is determined based on the time of removal of the last drain tube. The removal of the drain tube is assessed at the discretion of the surgeon.

CONTACTS AND LOCATIONS:
Overall Officials: Saleh K Saleh, MD, Principal Investigator — Minia University
Locations (1):
- Liver and GIT hospital / Minia university, Minya, Egypt

IPD SHARING:
Plan to Share IPD: No